CLINICAL TRIAL: NCT04025294
Title: The Evaluation of a School Climate Videogame Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000026033
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Reappraisal; Self Efficacy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Students playing videogame (Experimental): The experimental group will consist of our videogame intervention including the five mini-games.
  Interventions: Device: videogame
- Students receiving school climate assessment (Active Comparator): The control group differs from the experimental group as it includes the school climate assessment tool but excludes the mini-games
  Interventions: Behavioral: School Climate Assessment Survey

INTERVENTIONS:
Device: videogame — A videogame intervention that is interactive and engaging that teaches adolescents how to restructure negative automatic thoughts through an adapted thought record (a technique used in cognitive behavioral therapy to improve moods) by modeling how to do so and then empower them through real-life activities to improve their school climate. The videogame intervention is comprised of five mini-games, each containing a short narrative that models how to restructure negative automatic thoughts and navigate through challenging situations that often take place in school settings. The topics of each mini-game are informed by the constructs of school climate according to the National School Climate Center. Students using the videogame intervention will be prompted to think deeply and reflect on the narratives presented in each mini-game.
  Arms: Students playing videogame
Behavioral: School Climate Assessment Survey — A school climate assessment survey will include items adapted from questions developed by the National School Climate Center. Items will assess various dimensions of school climate including safety, social media, relationships, support for learning, and environment.
  Arms: Students receiving school climate assessment

SUMMARY:
A randomized control trial of a videogame intervention to assess and improve school climate.

DETAILED DESCRIPTION:
To assess the acceptability and preliminary efficacy of a videogame intervention designed to teach teens the skills in restructuring thoughts and then empowering them to take action and improve their school climate.

For this project, the play2PREVENT Lab aims to assess the acceptability and preliminary efficacy of a videogame intervention designed to teach teens the skills in restructuring thoughts and then empowering them to take action and improve their school climate. Program and school staff will enroll participants between the ages of 14-19 years old to play our videogame during their after school programs. Before and after gameplay, participants will answer assessment questions related to self-efficacy, cognitive reappraisal, and dimensions of school climate. Questions will also assess participants' feedback on the videogame. Students not randomly assigned to the videogame intervention will only respond to assessment questions. The data will be transmitted electronically via Qualtrics data collection platform to the Lab for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must be a current high school student
* English-speaking
* Willing to provide minor assent
* Willing to provide parental consent (if under 18 years old)
* Willing to play/use the game/tool for about 45 minutes to 1 hour after school
* Willing to answer questions about their experiences in playing the game, questions around school climate, and questions around self-efficacy on an iPad for about 30 minutes
* Willing to participate in an optional focus group for about 30 minutes

Exclusion Criteria:

* Those that do not meet the criteria above

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Measuring self-efficacy at baseline | baseline
  Participants will complete a pre-survey through a secured, data collection website (Qualtrics), before playing the videogame. Items from the general self-efficacy questionnaire will assess participants' self-efficacy at baseline. This scale uses a 5-point Likert response scale (1=Never, 2=Almost Never, 3=Sometimes, 4=Fairly Often, 5=Very Often). Total self-efficacy score ranges from 10-50.
Change in self-efficacy from baseline | immediately after playing the videogame
  Participants will complete a post-survey through a secured, data collection website (Qualtrics), immediately after playing the videogame. Items from the general self-efficacy questionnaire will assess participants' self-efficacy at baseline. This scale uses a 5-point Likert response scale (1=Never, 2=Almost Never, 3=Sometimes, 4=Fairly Often, 5=Very Often). Total self-efficacy score ranges from 10-50.
Measuring emotional self-efficacy at baseline | baseline
  Participants will complete a pre-survey through a secured, data collection website (Qualtrics), at baseline. Items from the Self-Efficacy Questionnaire for Children (SEQ-C) will assess participants' emotional self-efficacy immediately before playing the game. Each of the 6 items used in the study has to be scored on a 5-point scale with 1 = not at all and 5 = very well.
Change in emotional self-efficacy from baseline | immediately after playing the videogame
  Participants will complete a post-survey through a secured, data collection website (Qualtrics), at baseline. Items from the Self-Efficacy Questionnaire for Children (SEQ-C) will assess participants' emotional self-efficacy immediately after playing the game. Each of the 6 items used in the study has to be scored on a 5-point scale with 1 = not at all and 5 = very well.
Cognitive reappraisal scores at baseline | at baseline
  Participants will complete a pre-survey through a secured, data collection website (Qualtrics), at baseline.
  The ERQ-CA includes 6 items assessing participants' cognitive appraisal. The scale length ranges up to five points with the following options: 1) strongly disagree; 2) disagree, 3) half and half, 4) agree, 5) strongly agree. The range of scores for each scale was 6 to 30.
Cognitive reappraisal scores at baseline | immediately after playing the videogame
  Participants will complete a post-survey through a secured, data collection website (Qualtrics), immediately after playing the videogame. Items from the Emotional Regulation Questionnaire for Children and Adolescents (ERQ-CA) will assess participants' cognitive reappraisal immediately after playing the tool/game.
  The ERQ-CA includes 6 items assessing participants' cognitive appraisal. The scale length ranges up to five points with the following options: 1) strongly disagree; 2) disagree, 3) half and half, 4) agree, 5) strongly agree. The range of scores for each scale was 6 to 30.

SECONDARY OUTCOMES:
Gameplay post-assessment | immediately after playing the game
  Participants will complete a post-survey through a secured, data collection website (Qualtrics), immediately after playing the game. Twelve items will assess intervention experience and satisfaction from items designed by members of the study team (e.g., How likely do you think completing any of the activities will help you improve how you feel about yourself, others, or social situations? Response options include very likely, likely, might or might not, unlikely, very unlikely.) These questions are not part of a larger scale.
School Climate | Baseline
  Participants will complete a pre-survey through a secured, data collection website (Qualtrics), immediately before playing the videogame. Items from the National School Climate Center will be adapted and used to assess dimensions of participants' school climate, including safety, support for learning, environment, social media, and relationships. Response options include yes, no, not applicable. These questions are not part of a larger scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Fiellin, MD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Health & Learning Games, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fernandes CF, Deng Y, Tran AH, Hieftje KD, Boomer TMP, Taylor CK, Fiellin LE. A Pilot Randomized Controlled Trial to Evaluate a Cognitive Behavioral Videogame Intervention: empowerED. Games Health J. 2023 Feb;12(1):42-52. doi: 10.1089/g4h.2021.0118. Epub 2022 Nov 8. PMID 36350349